CLINICAL TRIAL: NCT07044336
Title: Puxitatug Samrotecan (AZD8205) Monotherapy vs Chemotherapy in B7-H4 Selected Advanced/Metastatic Endometrial Cancer Who Progressed On or After Platinum Based Chemotherapy and Anti-PD-1/Anti-PD-L1 Therapy (Bluestar-Endometrial01)
Brief Title: Puxitatug Samrotecan (AZD8205) Monotherapy vs Chemotherapy in B7-H4-selected Endometrial Cancer (Bluestar-Endometrial01)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D6900C00003; GOG-3110 (Other: Gynecologic Oncology Group Foundation); ENGOT-en28 (Other: European Network for Gynaecological Oncological Trial groups)
Record Dates: First submitted 2025-06-23; First posted 2025-06-30 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Endometrial Cancer; Malignant Solid Tumour
Keywords: Bluestar-Endometrial01; AZD8205; Puxitatug Samrotecan; Puxi-Sam; Platinum-based chemotherapy; B7-H4; advanced/metastatic; Endometrial Cancer; Anti-PD-1; Anti-PD-L1; antibody-drug conjugate; Topoisomerase 1 Inhibitors; uterine neoplasm; female urogenital neoplasm
MeSH Terms: conditions — Endometrial Neoplasms; Neoplasm Metastasis; Uterine Neoplasms | interventions — Doxorubicin; Paclitaxel

STUDY DESIGN:
Intervention Model Description: Single Open-Label
Who Masked: Outcomes Assessor
Masking Description: Open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Puxitatug Samrotecan (Experimental): Puxi-Sam IV (intravenous) Q3W .
  Interventions: Drug: Puxitatug Samrotecan
- Chemotherapy (Active Comparator): Physician's choice of chemotherapy
  Doxorubicin IV Q3W or Paclitaxel IV on Days 1, 8, and 15 in 28 day cycles.
  Interventions: Drug: Doxorubicin; Drug: Paclitaxel

INTERVENTIONS:
Drug: Puxitatug Samrotecan — 2.4 mg/kg on Day 1 Q3W Route of administration: IV infusion
  Other Names: Puxi-Sam
  Arms: Puxitatug Samrotecan
Drug: Doxorubicin — 60 mg/m2 on Day 1 Q3W Route of administration: IV
  Other Names: ADRIAMYCIN®
  Arms: Chemotherapy
Drug: Paclitaxel — 80 mg/m2 on Days 1, 8, and 15 in 28-day cycle Route of Administration: IV
  Other Names: TAXOL®
  Arms: Chemotherapy

SUMMARY:
This is a Phase III, 2-arm, randomized, open label, multicenter, global study assessing the efficacy and safety of puxitatug samrotecan compared to physician's choice of chemotherapy (doxorubicin or paclitaxel) in participants with B7-H4 selected advanced/metastatic EC that progressed following platinum based chemotherapy and anti-PD-1/anti-PD-L1 therapy.

DETAILED DESCRIPTION:
The target population of interest in this study is participants with B7-H4-selected advanced/metastatic EC who have progressed on or after platinum-based chemotherapy and anti-PD-1/anti-PD-L1 therapy, either separately or in combination and should have received no more than 2 prior lines of therapy in advanced/metastatic setting. Participants will be randomized in a 1:1 ratio to Puxi-Sam (arm A) or physician's choice of chemotherapy (arm B; doxorubicin or paclitaxel). The total study size will be approximately 700 eligible participants.

During the treatment period, participants will receive Puxi-Sam IV Day 1 Q3W (Arm A) or either doxorubicin treatment IV Day 1 Q3W or paclitaxel treatment IV on Days 1, 8, and 15 in 28-day cycle (Arm B).

This study aims to see if Puxi-Sam allows participants to live longer without their endometrial cancer getting worse, or simply to live longer, compared to participants receiving standard of care chemotherapy. This study is also looking to see how the treatment and the endometrial cancer affects participants' quality of life.

ELIGIBILITY:
The main inclusion criteria include but are not limited to the following:

* Histologically confirmed diagnosis of endometrial carcinoma or carcinosarcoma.
* Recurrent/metastatic EC ie, with radiological or objective evidence of recurrence or progression.
* Has received prior platinum-based chemotherapy and anti-programmed cell death 1 protein (PD-1)/anti- programmed cell death ligand 1 (PD-L1) therapy, either separately or in combination.
* A WHO/ECOG performance status of 0 or 1 at Screening.
* Has radiographically measurable disease by RECIST 1.1

The main exclusion criteria include but are not limited to the following:

* Had uterine sarcomas or uterine neuroendocrine carcinoma.
* Has had a recurrence of endometrial carcinoma or carcinosarcoma more than > 12 months after completing platinum-based therapy administered in the curative-intent setting without any additional platinum-based therapy received in the recurrent setting.
* Had previously received treatment with any therapy (approved or investigational) that contained a TOP1i including ADCs .
* Had previously received treatment with Puxi-Sam or another B7-H4 targeting agent.
* History of (non-infectious) ILD/pneumonitis that required steroids, has current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at screening.
* Has clinically severe pulmonary compromise resulting from intercurrent pulmonary illnesses.
* Active or previously documented autoimmune or inflammatory disorders

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 700 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2027-11-02 (Estimated); Study Completion 2028-04-03 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) for Arm A vs Arm B | Approximately 3 years
  PFS is defined as the time from randomization until progression per RECIST 1.1 as assessed by BICR or death due to any cause.
Overall survival (OS) for Arm A vs Arm B | Approximately 3 years
  OS is defined as the time from randomization until the date of death due to any cause.

SECONDARY OUTCOMES:
Assessment of Overall Response Rate (ORR) for Arm A vs Arm B | Approximately 3 years
  ORR is defined as the proportion of participants who have a response of CR or PR, as determined by BICR assessments, per RECIST 1.1.
Assessment of Duration of response (DoR) for Arm A vs Arm B | Approximately 3 years
  DoR will be defined as the time from the date of first documented response until the date of documented progression per RECIST 1.1 as assessed by BICR, or death due to any cause.
Assessment of progression-free survival 2 (PFS2) for Arm A vs Arm B | Approximately 3 years
  PFS2 will be defined as the time from randomization to the earliest of the progression event (following the initial Investigator-assessed progression), after first subsequent therapy, or death.
Time until first subsequent anticancer therapy after discontinuation of the randomized treatment, or death (TFST) for Arm A vs Arm B | Approximately 3 years
  TFST is defined as the time from randomization until the start date of the first subsequent anticancer therapy after discontinuation of the randomized treatment, or death due to any cause.
Time until the second subsequent anticancer therapy after discontinuation of the first subsequent treatment, or death (TSST) for Arm A vs Arm B | Approximately 3 years
  TSST is defined as the time from randomization until the start date of the second subsequent anticancer therapy after discontinuation of the first subsequent treatment, or death due to any cause.
Time until discontinuation of treatment for any reason, or death (TDT) for Arm A vs Arm B | Approximately 3 years
  TDT is defined as the time from randomization until discontinuation of treatment for any reason, including disease progression, toxicity, and death.
Worsening in endometrial symptoms for Arm A vs Arm B | Approximately 3 years
  Time to worsening is defined as time from date of randomization to the date of worsening while on treatment for endometrial symptoms, physical functioning, and health-related quality of life based on select items from the EORTC IL389.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Slomovitz, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Stephanie Gaillard, MD, PhD, Principal Investigator — Johns Hopkins University - Sidney Kimmel Comprehensive Cancer Center (SKCCC); Nicole Concin, Prof., Principal Investigator — Head of the Division of General Gynecology and Gynecologic Oncology at the Department of Obstetrics and Gynecology of MedUni Vienna and University
Locations (238):
- United States (54):
  - Research Site, Phoenix, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, La Jolla, California
  - Research Site, Los Angeles, California
  - Research Site, Orange, California
  - Research Site, Jupiter, Florida
  - Research Site, Miami, Florida
  - Research Site, Miami Beach, Florida
  - Research Site, Orlando, Florida
  - Research Site, Honolulu, Hawaii
  - Research Site, Chicago, Illinois
  - Research Site, Peoria, Illinois
  - Research Site, Urbana, Illinois
  - Research Site, Fort Wayne, Indiana
  - Research Site, Indianapolis, Indiana
  - Research Site, Scarborough, Maine
  - Research Site, Baltimore, Maryland
  - Research Site, Silver Spring, Maryland
  - Research Site, Ann Arbor, Michigan
  - Research Site, Detroit, Michigan
  - Research Site, Minneapolis, Minnesota
  - Research Site, Camden, New Jersey
  - Research Site, Paramus, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, Brooklyn, New York
  - Research Site, The Bronx, New York
  - Research Site, White Plains, New York
  - Research Site, Greenville, North Carolina
  - Research Site, Pinehurst, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Dayton, Ohio
  - Research Site, Hilliard, Ohio
  - Research Site, Sylvania, Ohio
  - Research Site, Bethlehem, Pennsylvania
  - Research Site, Hershey, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Willow Grove, Pennsylvania
  - Research Site, Sioux Falls, South Dakota
  - Research Site, Knoxville, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Houston, Texas
  - Research Site, Tyler, Texas
  - Research Site, Fairfax, Virginia
  - Research Site, Falls Church, Virginia
  - Research Site, Norfolk, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Roanoke, Virginia
  - Research Site, Kennewick, Washington
  - Research Site, Seattle, Washington
  - Research Site, Morgantown, West Virginia
  - Research Site, Waukesha, Wisconsin
- Argentina (8):
  - Research Site, Capital Federal
  - Research Site, Ciudad Autonoma Buenos Aires
  - Research Site, Ciudad de Buenos Aires
  - Research Site, Córdoba
  - Research Site, Cuidad Autónoma de Buenos Aire
  - Research Site, La Rioja
  - Research Site, Pergamino
  - Research Site, Viedma
- Australia (6):
  - Research Site, Malvern
  - Research Site, Melbourne
  - Research Site, Randwick
  - Research Site, St Leonards
  - Research Site, Subiaco
  - Research Site, Westmead
- Austria (3):
  - Research Site, Graz
  - Research Site, Innsbruck
  - Research Site, Vienna
- Belgium (7):
  - Research Site, Brussels
  - Research Site, Charleroi
  - Research Site, Edegem
  - Research Site, Ghent
  - Research Site, Leuven
  - Research Site, Liège
  - Research Site, Namur
- Brazil (13):
  - Research Site, Blumenau
  - Research Site, Curitiba
  - Research Site, Florianópolis
  - Research Site, Natal
  - Research Site, Porto Alegre
  - Research Site, Recife
  - Research Site, Rio de Janeiro
  - Research Site, Salvador
  - Research Site, São Caetano do Sul
  - Research Site, São Paulo
  - Research Site, Sorocaba
  - Research Site, Taubaté
  - Research Site, Teresina
- Canada (2):
  - Research Site, Edmonton, Alberta
  - Research Site, Montreal, Quebec
- China (21):
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Dalian
  - Research Site, Fuzhou
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Jinan
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Shenzhen
  - Research Site, Shijiazhuang
  - Research Site, Tianjin
  - Research Site, Wenzhou
  - Research Site, Wuhan
  - Research Site, Xi'an
  - Research Site, Zhengzhou
- Czechia (6):
  - Research Site, Brno
  - Research Site, Hradec Králové
  - Research Site, Nový Jičín
  - Research Site, Ostrava
  - Research Site, Prague
  - Research Site, V Uvalu 84
- Research Site, Herlev, Denmark
- Finland (3):
  - Research Site, Kuopio
  - Research Site, Tampere
  - Research Site, Turku
- France (16):
  - Research Site, Avignon
  - Research Site, Besançon
  - Research Site, Bordeaux
  - Research Site, Chambray-lès-Tours
  - Research Site, Cholet
  - Research Site, Créteil
  - Research Site, Grenoble
  - Research Site, Lille
  - Research Site, Limoges
  - Research Site, Lyon
  - Research Site, Nantes
  - Research Site, Nîmes
  - Research Site, Paris
  - Research Site, Plerin SUR MER
  - Research Site, Rennes
  - Research Site, Toulouse
- Georgia (2):
  - Research Site, Batumi
  - Research Site, Tbilisi
- Germany (15):
  - Research Site, Amberg
  - Research Site, Chemnitz
  - Research Site, Dresden
  - Research Site, Essen
  - Research Site, Frankfurt am Main
  - Research Site, Freiburg im Breisgau
  - Research Site, Hamburg
  - Research Site, Heidelberg
  - Research Site, Heilbronn
  - Research Site, Mainz
  - Research Site, Münster
  - Research Site, Paderborn
  - Research Site, Regensburg
  - Research Site, Schwäbisch Hall
  - Research Site, Witten
- Greece (2):
  - Research Site, Athens
  - Research Site, Thessaloniki
- Hungary (3):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Győr
- Israel (9):
  - Research Site, Ashdod
  - Research Site, Hadera
  - Research Site, Haifa
  - Research Site, Holon
  - Research Site, Jerusalem
  - Research Site, Nahariya
  - Research Site, Ramat Gan
  - Research Site, Safed
  - Research Site, Tel Aviv
- Italy (15):
  - Research Site, Alessandria
  - Research Site, Aviano
  - Research Site, Bologna
  - Research Site, Catania
  - Research Site, Florence
  - Research Site, Haifa
  - Research Site, Milan
  - Research Site, Monza
  - Research Site, Napoli
  - Research Site, Parma
  - Research Site, Pisa
  - Research Site, Ponderano
  - Research Site, Roma
  - Research Site, Torino
  - Research Site, Vicenza
- Japan (19):
  - Research Site, Chūōku
  - Research Site, Hidaka-shi
  - Research Site, Isehara-shi
  - Research Site, Kashiwa-shi
  - Research Site, Kōtoku
  - Research Site, Kurume-shi
  - Research Site, Matsuyama
  - Research Site, Minatoku
  - Research Site, Nagoya
  - Research Site, Niigata
  - Research Site, Okayama
  - Research Site, Osaka
  - Research Site, Sapporo
  - Research Site, Sendai
  - Research Site, Suita
  - Research Site, Sunto-gun
  - Research Site, Toon-Shi
  - Research Site, Tsu
  - Research Site, Yokohama
- Lithuania (2):
  - Research Site, Kaunas
  - Research Site, Vilnius
- Netherlands (2):
  - Research Site, Amsterdam
  - Research Site, Maastricht
- Poland (2):
  - Research Site, Lodz
  - Research Site, Siedlce
- Slovenia (2):
  - Research Site, Ljubljana
  - Research Site, Maribor
- South Korea (5):
  - Research Site, Goyang-si
  - Research Site, Gwangjin-gu
  - Research Site, Seoul
  - Research Site, Songpa-gu
  - Research Site, Suwon
- Spain (10):
  - Research Site, Badalona
  - Research Site, Barcelona
  - Research Site, Córdoba
  - Research Site, El Palmar (Murcia)
  - Research Site, Hospitalet DEL Llobregat
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Santiago de Compostela
  - Research Site, Seville
  - Research Site, Valencia
- Taiwan (4):
  - Research Site, New Taipei City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
- United Kingdom (6):
  - Research Site, Bebington
  - Research Site, Canterbury
  - Research Site, Derby
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Truro

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/